CLINICAL TRIAL: NCT01698866
Title: Evaluation of the Immune Response After Vaccination Against Hepatitis B in Patients With Indolent Lymphoproliferative Disorders With no Treatment.
Brief Title: Low Grade Lymphoma
Acronym: EVACC-B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-004968-30
Record Dates: First submitted 2012-08-16; First posted 2012-10-03 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Indolent Lymphoproliferative Disorders
Keywords: Low grade lymphoma; follicular lymphoma; indolent lymphoproliferative disorders; Vaccin GenHevac B Pasteur
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccin GenHevac B Pasteur (Experimental): vaccin GenHevac B Pasteur (Suspension for injection in pre-filled syringe / 20 μg microgram(s)Per day). In total, 3 injections at M0, M1 and M6
  Interventions: Biological: Vaccin GenHevac B Pasteur

INTERVENTIONS:
Biological: Vaccin GenHevac B Pasteur

SUMMARY:
The purpose of this study is to assess the seroconversion rate and the cellular immune response after vaccination against hepatitis B virus in patients with lymphoproliferative syndrome like chronic lymphocytic leukemia stade A and follicular lymphoma without of treatment criteria.

DETAILED DESCRIPTION:
Rituximab is a human-mouse chimeric monoclonal antibody that targets the B-cell CD20. It is an indispensible drug for the treatment of B-cell lymphoproliferative syndrome which induced immunosuppression. So, the infectious complications increase. Reactivation of hepatitis B virus is one such complication that can lead in asymptomatic hepatitis to death. Prevention of hepatitis B reactivation is recommended like using nucleoside analog for patients with chronic hepatitis B or occult hepatitis and vaccination against virus for seronegative patients. The published data about efficacy of hepatitis b vaccination in onco-haematology are rare. therefore, we carried out a prospective study to assess efficacy of hepatitis B vaccination in patients with lymphoproliferative disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Lymphoproliferative indolent type of stage A CLL or follicular lymphoma with low tumor burden
* No indication of chemotherapy during the seven months of the vaccination protocol.

HBV serology negative for HBsAg / Ab HBs / HBc Ab.

* No history of vaccination against hepatitis B.

Exclusion Criteria:

* Indication of immediate chemotherapy.
* At least one HBV positive serologic marker .
* History of vaccination against HBV.
* Known neurodegenerative disease.
* Pregnancy.
* Febrile infection untreated.
* Known allergy to any vaccine component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Describe the seroconversion rates at month 7 (M7) defined for a threshold of HBs Ab> 10 IU / L. | Month 7

SECONDARY OUTCOMES:
- Describe the seroconversion rate in month 2 (M2) defined for a threshold of HBs Ab> 10 IU / L. | Month 2
Describe the cellular immune response post vaccination at M2 and M7. | Month 2 and Month 7
To study the influence of age on the rate of seroconversion. | Month 0, Month 2 and Month 7
Describe vaccine-tolerance at M2 and M7. | Month 2 and Month 7
To study the influence of sex on the rate of seroconversion. | Month 0, Month 2 and Month 7
To study the influence of lymphocyte count on the rate of seroconversion. | Month 0, Month 2 and Month 7
To study the influence of total immunoglobulin on the rate of seroconversion. | Month 0, Month 2 and Month 7
To study the influence of immunoglobulin M on the rate of seroconversion. | Month 0, Month 2 and Month 7

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FEUGIER, MD, PhD, Principal Investigator — Pôle Hématologie CHU Nancy Brabois, CHU de Nancy, Vandoeuvre les Nancy, FRANCE
Locations (1):
- Pôle Hématologie CHU Nancy Brabois, Vandœuvre-lès-Nancy, France